CLINICAL TRIAL: NCT02627261
Title: Comparison of Three Methods to Evaluate Residual Disease in Multiple Myeloma
Brief Title: Multiple Myeloma Minimal Residual Disease
Acronym: MMRD
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Janssen, LP (Industry)
Responsible Party: Sponsor
Other Study IDs: 69HCL15_0316
Record Dates: First submitted 2015-12-04; First posted 2015-12-10 (Estimated); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
Keywords: residual disease
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — a gene sequencing technology will be used on bone marrow samples to detect residual disease
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with multiple myeloma: blood samples and bone marrow aspirates will be collected in patients at different time point
  Interventions: Biological: blood samples and bone marrow aspirates will be collected

INTERVENTIONS:
Biological: blood samples and bone marrow aspirates will be collected — Serial analysis will be performed at different time point in order to evaluate the presence or absence of residual disease after different treatment steps (before treatment, after induction, after intensification, after consolidation)

SUMMARY:
Three methods including flow cytometry, next generation sequencing and determination of circulating tumor cells will be performed at different time points in patients with previously undiagnosed multiple myeloma in order to determine the most sensitive method to detect residual disease

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* previously undiagnosed myeloma
* eligible for high dose therapy and bone marrow transplantation
* signed consent

Exclusion Criteria:

* ongoing therapy for another neoplasia
* Patients with other hematologic malignancies,
* patients deprived of liberty for administrative or judicial reasons
* previously treated for myeloma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will focus on adult patients with multiple myeloma and who will receive a treatment with high-dose melphalan and autologous bone marrow transplantation
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2018-09-02 (Actual)

PRIMARY OUTCOMES:
Quantification of residual disease | Residual disease is assessed up to 18 months after inclusion
  study the sensitivity of the method of quantification of circulating tumor cells compared to 2 others methods of detection

SECONDARY OUTCOMES:
kinetic of variation of the residual tumor cells detected by flow cytometry method | 18 months
  % positive cells in bone marrow sample
kinetic of variation of the residual tumor cells detected by new generation sequencing method | 18 months
  % positive in bone marrow sample
kinetic of variation of the circulating tumor cells | 18 months
  number of cells / mL of blood

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Huriez, Lille
  - Centre Hospitalier Universitaire Hôtel-Dieu de Nantes, Nantes
  - Centre Hospitalier Lyon Sud, Pierre Bénité

IPD SHARING:
Plan to Share IPD: No